CLINICAL TRIAL: NCT07216339
Title: Effect of Gamification on 6-Minute Walk Test Performance and Engagement in Pediatric Neuromuscular Patients
Brief Title: Gamification Effects on the 6-Minute Walk Test in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Toupin (Other)
Responsible Party: Sponsor-Investigator, David Toupin, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 103847
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Neuromuscular Diseases in Children
Keywords: Gamification; Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified test (Experimental): child carries a Radio-frequency identification (RFID) tag to scan at each lap, watching avatar level up.
  Interventions: Other: Gamified 6MWT
- Standard test (Active Comparator): no game; same verbal cue every minute
  Interventions: Other: Standard 6MWT

INTERVENTIONS:
Other: Standard 6MWT — ATS-standard instructions, no electronic system; Conducted in hallway measuring total length of 90ft (27.4 meters). Patients will walk down-and-back. A seated rest period of ≥10 min separates the two tests to minimize fatigue carry-over.
  Arms: Standard test
Other: Gamified 6MWT — identical course but child carries a RFID tag; at each lap the child taps an on an RFID reader, awarding a point and leveling-up an on-screen avatar; Conducted in hallway measuring total length of 90ft (27.4 meters). Patients will walk down-and-back.A seated rest period of ≥10 min separates the two tests to minimize fatigue carry-over.
  Arms: Gamified test

SUMMARY:
The goal of this study is to learn if adding a game to the 6-minute walk test for children with neuromuscular disorders will increase enjoyment and motivation to complete the test.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of, or active evaluation for, a neuromuscular disorder
* Able to ambulate (with or without usual orthoses/assistive device) sufficiently to attempt a 6-minute walk.
* Note: Acceptable if the patient needs to take breaks or sit during the test. Those unable to finish are counted as protocol deviations, not exclusions.
* Medically stable on the test day (no acute illness or recent surgery that would contraindicate moderate exercise).
* Child able to understand simple instructions in English and provide assent (if applicable based upon age and developmental level); parent/guardian able to provide consent in English.

Exclusion Criteria:

* Non-ambulatory or unsafe to attempt walking as judged by the treating physician.
* Severe cognitive/behavioral impairment that precludes following instructions.
* Acute cardiopulmonary, orthopedic, or other medical condition that makes walking unsafe on the test day.
* Non-English-speaking family (materials are available only in English for this pilot).
* Any child/parent who declines consent/assent or withdraws at any time.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6 minute walk distance | Baseline and post intervention (approximately 20 minutes)
  Participants will walk back and forth in the clinic hallway for 6 minutes and distance will be recorded in meters

SECONDARY OUTCOMES:
Change in Children's OMNI Rate of Perceived Exertion (RPE) Scale | Baseline and post intervention (approximately 20 minutes)
  The OMNI RPE scale is a visual and numerical tool from 0-10 that helps individuals subjectively gauge the intensity of walking or running activity, with 0 representing no effort and 10 being maximal exertion.
Change in Physical Activity Enjoyment Scale (PACES) | Baseline and post intervention (approximately 20 minutes)
  The Physical Activity Enjoyment Scale (PACES) consists of 8 questions scored on a scale from 1 to 7, with a maximum score of 56 and a minimum score of 8. Higher scores indicate greater enjoyment of physical activity.
Recruitment Rate | 9 months
  percent of eligible participants successfully recruited in the study
Test completion rate | 9 months
  number of walk tests successfully completed compared to overall number of walk tests

CONTACTS AND LOCATIONS:
Overall Officials: David N Toupin, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No